CLINICAL TRIAL: NCT00883623
Title: A Prospective Single Center Trial of Treatment With Lenalidomide-Melphalan-Dexamethasone in Patients With AL Amyloidosis
Brief Title: A Trial of Treatment With Lenalidomide-Melphalan-Dexamethasone in Patients With Primary (AL) Amyloidosis
Acronym: LEOMEX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Heidelberg University (Other)
Collaborators: Gesellschaft fur Medizinische Innovation - Hamatologie und Onkologie mbH (Other)
Responsible Party: Principal Investigator, Dr. Stefan Schönland, MD, Heidelberg University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-001405-41; GMIHO 005/2007 (191063)
Record Dates: First submitted 2009-04-15; First posted 2009-04-17 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Primary Amyloidosis
Keywords: AL-Amyloidosis; Lenalidomide
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment Arm (Experimental): Treatment Arm
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide — Up to 6 cycles of oral L-Mel-Dex, every 28 days Revlimid® 10 mg daily for 21 days, (add on therapy), Melphalan 0.15 mg/kg/day day 1-4, Dexamethasone 20 mg day 1-4
  Other Names: Revlimid

SUMMARY:
The treatment with oral melphalan and prednisone has been recommended as standard treatment of AL amyloidosis but the results are rather disappointing. Another therapeutic option is pulsed high-dose dexamethasone + melphalan (Mel-Dex) with more encouraging results regarding the achievement of a faster disease response and higher rates of haematological remission. In the last 5 - 10 years, promising treatment outcomes after therapy with high-dose melphalan and autologous stem cell support have been reported by several groups but only highly selected patients are eligible for this treatment. Lenalidomide has been shown to be effective in phase II and III trials in MM patients. Because of the relationship to MM, Lenalidomide is a promising therapeutic option also for patients with AL amyloidosis. The addition of Lenalidomide to Mel-Dex could improve rate of complete response (CR) and organ response in patients not eligible for or refused high-dose chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven systemic untreated AL amyloidosis requiring systemic chemotherapy
* Not eligible for or refused HDM
* Measurable plasma cell disease
* Life expectancy > 3 months
* WHO performance status < 3
* NYHA < stage IV
* Understand and voluntarily sign an informed consent form
* Laboratory test results within these ranges Absolute neutrophil count > 1.5 x 109/L Platelet count > 100 x 109/L Creatinine Clearance / MDRD > 40 ml/min Total bilirubin > 2,5 mg/dL
* Females of childbearing potential (FCBP) must agree to use two reliable forms of contraception simultaneously or to practice complete abstinence from heterosexual intercourse during the following time periods related to this study: 1) for at least 28 days before starting study drug; 2) while participating in the study; and 3) for at least 28 days after discontinuation from the study.

Exclusion Criteria:

* Multiple Myeloma stage II and III (Durie and Salmon)
* Previous organ transplantation
* Not able to visit the Amyloid Clinic in Heidelberg once per month
* Refusal of aspiration of 100 ml bone marrow at study inclusion
* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
* Pregnant or breast feeding females. (Lactating females must agree not to breast feed while taking lenalidomide).
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
* Use of any other experimental drug or therapy within 28 days of baseline.
* Known hypersensitivity to thalidomide.
* The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
* Any prior use of lenalidomide.
* Concurrent use of other anti-cancer agents or treatments.
* Known positive for HIV or infectious hepatitis, B or C.
* Patients who are in a depending position of the Sponsor or the Principal Investigator

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-04; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Complete response (CR) rate | 6 months: after 6 cycles of L-Mel-Dex

SECONDARY OUTCOMES:
Rate of hematological response (CR and PR) | 6 months
Organ response rate | 3 months after discontinuation of L-Mel_Dex (maximum: 9 months)
Correlation of cytogenetic aberrations and gene expression profiling (GEP) results with best hematological response to treatment | 6 months
Retrospective comparison with a historical control group treated with Mel-Dex in our institution | 01.04.2012
Toxicity (hematological and non-hematological) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Schoenland, MD, Principal Investigator — University Clinic Heidelberg - Department of Internal Medicine V
Locations (1):
- University Clinic Heidelberg, Heidelberg, Germany

REFERENCES:
- [Derived] Hegenbart U, Bochtler T, Benner A, Becker N, Kimmich C, Kristen AV, Beimler J, Hund E, Zorn M, Freiberger A, Gawlik M, Goldschmidt H, Hose D, Jauch A, Ho AD, Schonland SO. Lenalidomide/melphalan/dexamethasone in newly diagnosed patients with immunoglobulin light chain amyloidosis: results of a prospective phase 2 study with long-term follow up. Haematologica. 2017 Aug;102(8):1424-1431. doi: 10.3324/haematol.2016.163246. Epub 2017 May 18. PMID 28522573